CLINICAL TRIAL: NCT00736528
Title: An Investigator And Subject-Blind, Phase 1 Study To Characterize The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Multiple Doses Of PF-04447943 In Healthy Elderly Subjects
Brief Title: A Phase I, Multiple Dose Study of PF-04447943 in Healthy Elderly Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See Detailed Description for termination reason.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B0401002
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Healthy; Elderly
Keywords: safety, tolerability, pharmacokinetics, cognition
MeSH Terms: interventions — 6-(4-methyl-1-(pyrimidin-2-ylmethyl)pyrrolidin-3-yl)-1-(tetrahydro-2H-pyran-4-yl)-1,5-dihydro-4H-pyrazolo(3,4-d)pyrimidin-4-one

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-04447943 05 mg dose (Experimental)
  Interventions: Drug: PF-04447943
- PF-04447943 15 mg dose (Experimental)
  Interventions: Drug: PF-04447943
- PF-04447943 45 mg dose (Experimental)
  Interventions: Drug: PF-04447943
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04447943 — 05 mg BID for 14 days
  Arms: PF-04447943 05 mg dose
Drug: PF-04447943 — 15 mg BID for 14 days
  Arms: PF-04447943 15 mg dose
Drug: PF-04447943 — 45mg BID for 14 days
  Arms: PF-04447943 45 mg dose
Drug: Placebo — Placebo for 14 days
  Arms: Placebo

SUMMARY:
To describe the safety, tolerability and pharmacokinetics of PF-04447943 after administration of multiple, ascending, oral doses to healthy elderly subjects.

DETAILED DESCRIPTION:
Additional Study Purpose Details: Phase I safety and pharmacokinetics study.

Detailed Description:

The study was terminated on 11/12/2008. There were no safety findings in this trial that resulted in the decision to terminate the trial. The study was closed in order to change the amount of drug that subjects would take and to shorten the number of days that the drug would be taken in a new study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Elderly
* 65-85

Exclusion Criteria:

* Evidence or history of clinically significant unstable disease

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Primary Safety: Adverse events, change from baseline in vital signs, triplicate ECG, clinical safety laboratory endpoints | 14 days
Pharmacokinetic endpoints will include plasma PF 04447943 AUCt, Cmax and Tmax | 14 days

SECONDARY OUTCOMES:
Changes in cognition from baseline | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Gainesville, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0401002&StudyName=A%20phase%20I%2C%20multiple%20dose%20study%20of%20PF-04447943%20in%20healthy%20elderly%20volunteers